CLINICAL TRIAL: NCT06420453
Title: How Long Can Labor Last? Person Centred Care During Labor to Increase Safety for Women and Newborn
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Mia Ahlberg, Associate Professor, Karolinska Institutet
Other Study IDs: 2023-02010
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Birth Outcome, Adverse; Labor Long; Labor Complication; Maternal Injury; Maternal Distress During Labor and Delivery; Neonatal and Perinatal Conditions; Labor Duration
MeSH Terms: conditions — Pregnancy Complications; Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed to prolonged labor duration
- Not exposed to prolonged labor duration

SUMMARY:
"How long will my labor last" is a very common question for midwives who care for women during birth. To evaluate safe labor duration largely determines management and care during birth. Today a standardized tool is used by midwives to evaluate normal and safe labor called the partograph. The World Health Organization partograph is a decision-making support tool designed to assist midwives in identifying normal labor duration and women at risk of developing complications. The tool guide the use of care interventions intended to mitigate any perceived risks. The partograph has been in use since the 1950ies and has had a profound impact on care and management during labor. Normal labor progression according to the partograph is a linear progression with cervical dilation of 1 centimeter per hour (alert line) and any deviation from this should lead to an intervention.The purpose of this research project is to increase person-centred care during labor. Specifically, we want to provide updated comprehensive information on labor duration and patient safety for reduction of; unnecessary medical interventions during normal labor; morbidity and mortality in the new-born; maternal complications during delivery and the puerperal period.

ELIGIBILITY:
Inclusion Criteria:

All births with labor duration

Exclusion Criteria:

Elective Cesarean birth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an epidemiological research project using the largest cohort in the world containing detailed information on labor progression and care during labor. The cohort used is built from detailed data from medical records in the Stockholm-Gotland Obstetric Cohort, including all births from 2008 to 2020 (> 300 000 births). This includes data from the partograph with information about start of labor, all cervical examinations, care interventions, total duration of labor, maternal and neonatal outcomes. For completeness of data on infant outcomes, the cohort has been linked with the Swedish Neonatal Quality Register (SNQ).
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse neonatal outcomes | 1 month postpartum
Adverse maternal outcomes | 1 month postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No